CLINICAL TRIAL: NCT02473731
Title: A Window of Opportunity Study of KTN3379 in Surgically Resectable Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTN3379-CL-002
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2017-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: CDX3379
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Treatment with KTN3379 in HPV positive head and neck cancer patients
  Interventions: Biological: KTN3379
- B (Experimental): Treatment with KTN3379 in HPV negative head and neck cancer patients
  Interventions: Biological: KTN3379

INTERVENTIONS:
Biological: KTN3379

SUMMARY:
The purpose of this study is to evaluate the activity and safety of KTN3379 in head and neck cancer patients and to explore downstream molecular pathways to identify tumor response and resistance mechanisms by evaluating various biomarkers before and after treatment.

DETAILED DESCRIPTION:
This is an open-label study in patients with squamous cell carcinoma of the head and neck (SCCHN) scheduled for surgery. Two cohorts of SCCHN patients, HPV negative and HPV positive, will be treated with KTN3379 to evaluate effects on ErbB3 phosphorylation and other biomarkers in tumor tissue. The KTN3379 treatment duration is within the expected window of time that elapses from initial patient evaluation by a surgeon to performance of surgery. Paired preoperative and postoperative tumor specimen analyses allow evaluation of proliferation, ErbB3 related biomarkers, pErbB3 modulation and pharmacodynamic changes in downstream molecular pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed primary, untreated SCCHN including variants. Patients must be candidates for surgical resection. Primary tumors of oral cavity, oropharynx, hypopharnyx or larynx are included.
2. Written informed consent and any locally required authorization (e.g., HIPAA in the USA) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
3. Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for 60 days after the final dose of KTN3379. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are postmenopausal (defined as 12 months with no menses without an alternative medical cause)
4. Nonsterilized males who are sexually active with a female partner of child-bearing potential must, with their partner, use 2 acceptable methods of effective contraception from Day 1 through 60 days after receipt of the final dose of KTN3379.
5. Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
6. Adequate bone and marrow function as defined below:

   * Hemoglobin ≥ 10 g/dL
   * Absolute neutrophil count ≥ 1500/mm3
   * Platelet count ≥ 100,000/mm3
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ×ULN
   * Bilirubin ≤ 1.5 × ULN except for cases of documented or suspected Gilbert's disease, in which bilirubin must be ≤ 5 × ULN
   * Serum creatinine ≤ 1.5 g/dL
   * Normal PT or INR and aPTT

Exclusion Criteria:

1. Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
2. Immunosuppressive or systemic steroids medication within 7 days before the first dose of KTN3379 (inhaled and topical corticosteroids are permitted).
3. Another invasive malignancy within 2 years prior to enrollment except for localized prostate cancer, cervical carcinoma in situ, non-melanomatous carcinoma of the skin, or ductal carcinoma in situ of the breast that has/have been surgically cured
4. Major surgical procedure within 30 days prior to Day 1 or incomplete recovery from any prior surgery
5. Pregnancy or lactation
6. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled or idiopathic hypotension, unstable angina pectoris, cardiac arrhythmia including atrial fibrillation, significant cardiac conduction abnormalities including prolongation of QTc interval or BBB, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
7. Patients with a left ventricular cardiac ejection fraction < 50% as assessed by an echocardiogram or MUGA scan
8. Patients with prior primary treatment for head and neck cancer (e.g. chemoradiation or radiation alone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Change in pErbB3 levels in tumor tissue | 4 weeks
  Reduction in pErbB3 levels

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 6 weeks
  Adverse events (AEs), serious adverse events (SAEs), laboratory evaluations, radiological assessments, vital signs, electrocardiograms (ECGs), and physical examinations.
Ki67 proliferative index in tumor tissue | 4 weeks
  Ki67 proliferative index in tumor tissue before and after treatment
Changes in tumor measurements (RECIST 1.1 measurements) | 4 weeks
  RECIST 1.1 measurements before and after treatment
Pharmacokinetics (Peak plasma concentrations of KTN3379 Trough plasma concentrations of KTN3379) | 4 weeks
  Peak plasma concentrations of KTN3379 Trough plasma concentrations of KTN3379
Anti drug antibodies | 6 weeks
  Measurement of anti KTN3379 antibodies in blood

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Duvvuri U, George J, Kim S, Alvarado D, Neumeister VM, Chenna A, Gedrich R, Hawthorne T, LaVallee T, Grandis JR, Bauman JE. Molecular and Clinical Activity of CDX-3379, an Anti-ErbB3 Monoclonal Antibody, in Head and Neck Squamous Cell Carcinoma Patients. Clin Cancer Res. 2019 Oct 1;25(19):5752-5758. doi: 10.1158/1078-0432.CCR-18-3453. Epub 2019 Jul 15. PMID 31308059